CLINICAL TRIAL: NCT06531694
Title: Unravelling the Interplay of Weight Stigma and Pregnancy Outcomes: A Prospective Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Monash University (Other)
Responsible Party: Sponsor
Other Study IDs: 601966989
Record Dates: First submitted 2024-07-07; First posted 2024-08-01 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Weight Stigma; Pregnancy Outcomes; Overweight and Obesity
Keywords: Prenatal care; Healthcare
MeSH Terms: conditions — Weight Prejudice; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective cohort study is to investigate the contribution of stigma and discrimination due to body size to adverse pregnancy outcomes. We also aim to explore the role of psychological and social factors in this relationship. The specific objectives of this study are:

Objective 1: Explore weight stigma as a mediator of the association between BMI ≥30 kg/m2 and adverse pregnancy outcomes.

Objective 2: Explore confounding factors not previously considered such as weight cycling, trauma, eating disorders, and internalised weight bias as mediators in the relationship between obesity and adverse pregnancy outcomes.

DETAILED DESCRIPTION:
The specific research questions for each objective are:

Objective 1 RQ1.1: Does weight stigma experienced during pregnancy in a healthcare setting reported up to 34 weeks gestation mediate the association between pre-pregnancy obesity (BMI ≥30) and gestational diabetes mellitis (GDM) (primary outcome)?

RQ1.2: Does weight stigma experienced during pregnancy in a healthcare setting reported up to 34 weeks gestation mediate the association between pre-pregnancy obesity (BMI ≥30) and (i) induction of labour; (iv) mode of birth; (ii) gestational hypertension (any); (iii) infant birth weight; and (iv) establishment of breastfeeding by 6 weeks postpartum (secondary outcomes)?

Objective 2:

RQ2.1: Do weight cycling, history of trauma, history of eating disorders, and internalised weight bias explain any of the variance in the mediation relationships described above?

ELIGIBILITY:
Inclusion Criteria:

* Pregnant between 10-22 weeks' gestation
* Greater or equal than 18 years of age
* Booked to give birth at Adelaide Women's and Children's Hospital or Royal Women's and Children's Brisbane
* Access to the Internet to complete the survey
* Consents to the extraction of hospital electronic medical record data about the woman and relevant to the study.
* Ability to read and understand English

Exclusion Criteria:

* Pregnant with multiple gestation
* Insufficient English language skills to consent and complete the questionnaires.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who are pregnant between 10-22 weeks gestation
Study Population: Participants will be pregnant women who are at least 18 years old with a singleton pregnancy, and who are booked in to give birth at Adelaide Women's and Children's Hospital or Royal Women's and Children's Brisbane. At baseline, women must be between 10 and 22 weeks' gestation.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of women diagnosed with gestational diabetes mellitis by 34 weeks gestation | 34 weeks
  Measuring the number of women reporting a diagnosis of gestational diabetes mellitis by 34 weeks gestation as assessed via self-reported measures and chart review.

SECONDARY OUTCOMES:
Proportion of women experiencing induction of labour | 6 weeks postpartum
  Identifying whether the woman's labour was spontaneous or induced measured via a self-reported questionnaire.
Proportion of women reporting each mode of birth (i.e., vaginal birth, caesarean section, assisted vaginal birth, or other) | 6 weeks postpartum
  Identifying the mode of birth assessed via a self-reported questionnaire. Options are: vaginal birth, caesarean section, assisted vaginal birth (e.g., with forceps), or other.
Proportion of women who reported experiencing gestational hypertension in their most recent pregnancy | 6 weeks postpartum
  Identifying the proportion of women who reported a diagnosis of gestational hypertension during their most recent pregnancy via a self-reported questionnaire.
Infant birth weight (in grams) reported by mothers for their most recent infant | 6 weeks postpartum
  Infant birth weight (in grams) reported by mothers based on their most recent baby's birth certificate or hospital discharge summary information.
Proportion of women currently breastfeeding their infant reported by mothers at 6-weeks postpartum | 6 weeks postpartum
  The proportion of women currently breastfeeding their infant (yes/no) reported by mothers at 6-weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Briony Hill, PhD, Principal Investigator — Monash University